CLINICAL TRIAL: NCT01857453
Title: National, Multicentric, Prospective Phase II Study Estimating the Interest of a Dose Decrease for Radiation Therapy Associated With a Carboplatine and Etoposide Based Chemotherapy for the Treatment of Standard Risk Adult Medulloblastomas
Brief Title: Interest of a Dose Decrease for Radiotherapy Associated With Chemotherapy for Treatment of Standard Risk Adult Medulloblastomas
Acronym: RSMA2010
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Bordeaux (Other); Centre Paul Strauss (Other); Centre Hospitalier Universitaire de Nice (Other); CRLCC Val d'Aurelle, Montpellier (Unknown); Centre Georges Francois Leclerc (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Centre Leon Berard (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Hôpital de la Timone (Other); CHU de Reims (Other); Hopitaux Civils de Colmar (Other); University Hospital, Lille (Other); Institut Claudius Regaud (Other); Centre Francois Baclesse (Other); Center Eugene Marquis (Other); Centre René Gauducheau (Other); Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-002803-16
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Medulloblastoma
Keywords: Adult Patients Medulloblatoma Standard risk group Chemotherapy Radiotherapy Quality of Life
MeSH Terms: conditions — Medulloblastoma | interventions — Carboplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- teatment arm (Experimental): carboplatine + etoposide based chemotherapy followed by radiation therapy with 24 Gy on the in toto neuro axis and 54 Gy on the post operative bed
  Interventions: Drug: carboplatine; Drug: Etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatine — carboplatine + etoposide based chemotherapy followed by radiation therapy with 24 Gy on the in toto neuro axis and 54 Gy on the post operative bed
Drug: Etoposide — carboplatine + etoposide based chemotherapy followed by radiation therapy with 24 Gy on the in toto neuro axis and 54 Gy on the post operative bed
Radiation: radiation therapy — carboplatine + etoposide based chemotherapy followed by radiation therapy with 24 Gy on the in toto neuro axis and 54 Gy on the post operative bed

SUMMARY:
Adult medulloblastoma is a rare tumour.

The "standard risk " group (complete surgery or residual tumour lower than 1,5 cm2, absence of malignant cells in the cerebrospinal fluid, absence of metastasis, absence of MYC amplification and exclusion of large cells medulloblastoma) concerns, for the adult population, a majority of patients at diagnosis (about ¾ of cases).

Conventional treatment is classically based on a 54/36 Gy cranio-spinal radiotherapy (54 Gy on the posterior fossa and 36 Gy on the nevraxis).

This treatment is associated with an acute toxicity (haematological, cutaneous, digestive and general) wich decreases gradually when patient goes away from the treatment period.

For this category of patients and this modality of treatment, The French intergroup experience, pleads in favour of a late and progressive neurotoxicity.

This neurotoxicity is associated with a clear degradation of the quality of life.

In the light of paediatric studies :

We propose a phase II study to estimate the interest of a decrease of radiation doses compensated by a chemotherapy according to the following schedule

1. carboplatine + etoposide based chemotherapy every 28 days x 2
2. followed by, less than 80 days after the surgery, radiation therapy with 24 Gy on the in toto neuro axis and 54 Gy on the post operative bed.

The majority of French centres concerned with the neuro-oncology are involved in this trial.

About 25 new cases by year are waited. A centralized analysis of pathological slides and of the pre and post surgery Magnetic Resonance Imaging is foreseen.

The main objective is to estimate the survival without disease at 1 year

Secondary objectives associate the evaluations of the rate of complete response at the end of procedure, the overall survival, the survival without disease, the survival without events, the neurocognitiv toxicity, the endocrine toxicity, the hearing toxicity and the time until definitive deterioration of the quality of life Associated studies

Two associated studies are besides foreseen (parallel search for co-financing):

1. A biologic study is planed with the aim to confirm, by morphological, genomic and transcriptomic studies, the interest, for the adult population, of the prognostic markers used in paediatric population
2. A radiological study is planed with the aim to estimate the interest :

   * of a multimodal follow-up (spectroscopy and perfusion imaging) for the premature detection of recurrences
   * of the study of functional connectivity in correlation with the neuropsychological follow-up for the analysis of the aetiology and premature markers of neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of medulloblastoma expect large cells type
* Patients between 18 and 70 years
* Résidual tumor les than 1.5 square centimeter (greater diameter)
* No sus tentorial or spinal location
* Absence of tumoral cells in the cerebrospinal fluid taken before, during or 14 days after surgery
* Absence of MYC amplification
* AID, B and C hepatitis positive serologies
* Negative βHCG dosage and effective contraception for potentially pregnant women
* Writed consent obtain

Exclusion Criteria:

* Age < 18 or > 70 years
* Previous diagnosis of medulloblastoma
* Previous treatment with chemotherapy
* Previous cranial or spinal radiation therapy
* Carboplatinum or etoposide contraindication
* Previous cancer in the five years before the inclusion except basocellular carcinoma of the skin and in situ cancer of the uterine cervix
* Severe renal renal insufficiency with a creatinine clearance < 60 ml/min
* Liver insufficiency with a contraindication of carboplatinum or etoposide based chemotherapy or elevated transaminases > 3N.
* Insufficient haematopoetic reserve (thrombocytes < 100 000/mm3 ou neutrophil polynuclear < 1500/mm3)
* Previous organ transplantation or immunosuppression
* Pregnant women or women without contraception
* Incapacity of respecting the recommanded follow up
* Participation in another therapeutic clinical trial
* Patient under custody
* Not social security regime membership

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2013-04-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
survival without disease at 1 year | one year

CONTACTS AND LOCATIONS:
Overall Officials: Luc TAILLANDIER, Principal Investigator — CHU NANCY - France
Locations (20):
- France (20):
  - Chu Amiens, Amiens
  - Chu Bordeaux, Bordeaux
  - CHU CAEN, Caen
  - Hopitaux Civils de Colmar, Colmar
  - Cenre Georges Francois Leclerc, Dijon
  - Chru de Lille, Lille
  - Centre Leon Berrard, Lyon
  - Hopital de La Timone, Marseille
  - Centre Val D'Aurelle, Montpellier
  - Chu Nancy, Nancy
  - Centre René Ganducheau, Nantes
  - Chu de Nice, Nice
  - Chu Nimes, Nîmes
  - Institut Curie, Paris
  - AP HP Groupe Hospitalier Pitié Salpétrière, Paris
  - Institut du Cancer COURLANCY, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Paul Strauss, Strasbourg
  - Chu de Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif